CLINICAL TRIAL: NCT06630507
Title: Measuring Change in Overcoming Implicit Biases in Behavior by Emergency Care Center Providers
Status: Not yet recruiting | Type: Observational
Sponsor: Sarasota Memorial Health Care System (Other)
Responsible Party: Principal Investigator, Katie West, MSN, RN, CEN, Sarasota Memorial Health Care System
Other Study IDs: 23-MEDI-99
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Implicit Bias
Keywords: healthcare providers; implicit bias; emergency care center
MeSH Terms: conditions — Bias, Implicit

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECC staff receiving educational module: Active healthcare providers (including emergency medicine physicians, nurse practitioners, physician assistants, and residents, as well as nurses, multi-skilled technicians, and paramedics) in the SMH-Sarasota ECC will fill out the initial surveys, complete the implicit bias education, and do the posttest (re-administer the Measuring Change in Overcoming Implicit Biases in Behavior by Emergency Medicine Personnel questionnaire).
  Interventions: Behavioral: Educational module
- ECC staff not receiving educational module: Active healthcare providers (including emergency medicine physicians, nurse practitioners, physician assistants, and residents, as well as nurses, multi-skilled technicians, and paramedics) in the SMH-Venice ECC will fill out the initial surveys and do the posttest (re-administer the Measuring Change in Overcoming Implicit Biases in Behavior by Emergency Medicine Personnel questionnaire).
  Once all data is collected from both groups, the Venice Campus ECC will be given the ECC implicit bias education.

INTERVENTIONS:
Behavioral: Educational module — 1 hour pre-recorded educational module created by Dr. Sharma.
  Groups: ECC staff receiving educational module

SUMMARY:
Implicit bias is a form of bias in which a person's automatic and unintentional thoughts of another person or group influence either positively or negatively their behavior or the decisions they make. Studies show that healthcare providers have the same amount of bias as any other person and that it can affect patient care. However, in the emergency room, which is fast-paced and there is a high number of patients, implicit bias may be higher. Therefore, this study will look at emergency care center (ECC) providers' willingness to change their implicit bias behaviors. After, it will provide implicit bias education designed for the ECC to the healthcare providers at SMHCS Sarasota campus and assess whether it improved their willingness to change implicit bias behaviors when compared to the providers in the SMHCS Venice campus who did not receive the education.

DETAILED DESCRIPTION:
Studies have shown that implicit bias is present in healthcare providers, including those in the emergency room, it is necessary to understand whether emergency providers are willing to change their implicit bias behaviors and provide them with the education and resources tailored to it so that they can be aware of it and make a positive change towards improving it even when they are pressured by time and never-ending tasks.

The observational study will use a two-group pretest-posttest design to assess willingness to change implicit bias behaviors among healthcare staff in the ECC. Healthcare providers will be recruited from two SMHCS clinical sites: Sarasota Memorial Hospital's (SMH) -Sarasota Campus ECC and SMH's-Venice Campus ECC.

Participants are expected to fill out the initial surveys, complete the implicit bias education, and do the posttest (re-administer the Measuring Change in Overcoming Implicit Biases in Behavior by Emergency Medicine Personnel questionnaire), which is expected to take approximately 6-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be eligible for the study if they are 18 years or older and are active emergency medicine staff in the SMH-Sarasota or the SMH-Venice campus ECC. Participants must also be able to understand the requirements of the study, be willing and able to provide informed consent, and participate in all required study activities.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare providers (including emergency medicine physicians, nurse practitioners, physician assistants, and residents, as well as nurses, multi-skilled technicians, and paramedics) from Sarasota Memorial Health Care System's two emergency care centers, Sarasota and Venice campuses.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Examine emergency care center (ECC) staff's willingness to overcome pre-existing implicit bias. | 6-18 months
  Administer the Measuring Change in Overcoming Implicit Biases in Behavior by Emergency Medicine Personnel questionnaire and asses scores.
Assess whether an educational module on implicit bias designed explicitly for the ECC increases willingness to overcome implicit bias behavior among ECC staff. | 6-18 months
  Administer the Measuring Change in Overcoming Implicit Biases in Behavior by Emergency Medicine Personnel questionnaire and assess scores.
Compare willingness to overcome implicit bias in ECC staff who received education versus staff who were not provided with any education. | 6-18 months
  Administer the Measuring Change in Overcoming Implicit Biases in Behavior by Emergency Medicine Personnel questionnaire and compare to the ECC staff who did not receive the education's scores.

CONTACTS AND LOCATIONS:
Overall Officials: Katie West, MSN, RN, CEN, Principal Investigator — Sarasota Memorial Health Care System
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brockett-Walker C, Lall M, Evans DD, Heron S. Racial Bias Among Emergency Providers: Strategies to Mitigate Its Adverse Effects. Adv Emerg Nurs J. 2021 Apr-Jun 01;43(2):89-101. doi: 10.1097/TME.0000000000000352. PMID 33915556
- [Background] FitzGerald C, Hurst S. Implicit bias in healthcare professionals: a systematic review. BMC Med Ethics. 2017 Mar 1;18(1):19. doi: 10.1186/s12910-017-0179-8. PMID 28249596
- [Background] Narayan MC. CE: Addressing Implicit Bias in Nursing: A Review. Am J Nurs. 2019 Jul;119(7):36-43. doi: 10.1097/01.NAJ.0000569340.27659.5a. PMID 31180913
- [Background] Shah HS, Bohlen J. Implicit Bias. 2023 Mar 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK589697/ PMID 36944001
- [Background] Thirsk LM, Panchuk JT, Stahlke S, Hagtvedt R. Cognitive and implicit biases in nurses' judgment and decision-making: A scoping review. Int J Nurs Stud. 2022 Sep;133:104284. doi: 10.1016/j.ijnurstu.2022.104284. Epub 2022 May 24. PMID 35696809